CLINICAL TRIAL: NCT01130207
Title: Effects of Bariatric Surgery on the Gastro-intestinal Microflora
Brief Title: Microbes and Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Edward J. Shillitoe, Professor, State University of New York - Upstate Medical University
Other Study IDs: Microbes and Bariatric Surgery
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Obesity; Diabetes; Periodontal Disease
Keywords: Obesity; Diabetes; Periodontal disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial samples from dental plaque and feces, and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will study people who are obese and will be treated by bariatric surgery. The investigators will test the hypothesis that some of the features of obesity are related to the bacteria in the gastro-intestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Will undergo bariatric surgery for treatment of obesity in Syracuse NY
* Willingness to participate

Exclusion Criteria:

* Any previous gastrointestinal surgery
* Use of antibiotics in the previous 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity who are already accepted for treatment by bariatric surgery in Syracuse NY
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in microflora after bariatric surgery | Six months
  Specific differences were measured in oral and intestinal bacteria immediately after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Upstate Medical University, Syracuse, New York, United States